CLINICAL TRIAL: NCT04258566
Title: A Feasibility Study to Evaluate the Combination of Electromagnetic Tracking and Optical Imaging With Indocyanine Green (ICG) for Hepatic Biopsies
Brief Title: Electromagnetic Tracking and Optical Imaging With ICG for Hepatic Biopsies
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulty
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 200039; 20-CC-0039
Record Dates: First submitted 2020-02-05; First posted 2020-02-06 (Actual); Results first posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatic Carcinoma; Indocyanine Green (ICG); Optical Imaging
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Optical plus fusion for liver biopsy (Experimental): Participants with diagnosed or suspected hepatocellular carcinoma (HCC) or metastatic intrahepatic cancer have the optical molecular imaging (OMI) performed with electromagnetic (EM) tracking during liver biopsy. Participants receive Indocyanine Green (ICG) 0.5 mg/kg, up to 40mg, intravenously 18-24hrs prior to scheduled biopsy.
  Interventions: Device: Optical Molecular Imaging (OMI); Radiation: Indocyanine Green (ICG); Device: Electromagnetic Tracking

INTERVENTIONS:
Device: Optical Molecular Imaging (OMI) — Tracks and localizes intrahepatic lesions
Radiation: Indocyanine Green (ICG) — Fluorescent dye used for visualization of cells and tissue
Device: Electromagnetic Tracking — Tracks and localizes intrahepatic lesions

SUMMARY:
Background:

Liver cancer is the sixth most common cancer worldwide. Diagnosing liver cancer usually requires a liver sample. Getting the best sample helps determine whether cancer is present and what kind of cancer it is. But sampling can be difficult. This study will look at combining two devices to provide better liver samples.

Objective:

To see if combining fusion imaging and optical imaging can better sample areas of concern in the liver and determine the presence of disease.

Eligibility:

People ages 18 and older who need a liver biopsy as part of diagnosis or treatment.

Design:

Participants will be screened with:

* Review of imaging
* Medical history
* Physical exam
* Blood test results

Participants will have a dye injected into a vein 24 hours before their biopsy. They will be monitored for 30 minutes for any side effects.

For the biopsy, participants skin will be numbed. They may have stickers placed on their belly to help guide the needle. They will have a CT scan to plan the needle s pathway. For the scan, they will lie in a machine that takes pictures of the body. A small camera will be placed near the needle to take pictures of the liver. A medical global positioning system (GPS) tracking system will be used. This will guide the needle into the area of the participant s liver where the biopsy will be taken.

After the biopsy, participants will recover in the hospital for 4 6 hours.

After the procedure, researchers will take the participants biopsy tissue and look at it to try to compare new ways to picture the sample.

DETAILED DESCRIPTION:
* Pilot study to evaluate the combination of optical molecular imaging (OMI) and EM tracking in localizing intrahepatic lesions and assess the concordance between fluorescence ICG and histopathology for the diagnosis of liver cancer.
* Hepatocellular Carcinoma (HCC) is the 3rd most common cause of cancer globally with an increasing incidence worldwide. Percutaneous sampling of focal hepatic lesions is a cornerstone in management of patients with hepatic pathology. In a retrospective study of patients with small hepatic lesions, up to 45% of the lesions biopsied were insufficiently visualized and resulted to a false negative rate (defined as patients with benign biopsies who were subsequently found to have malignant lesions at the attempted site of biopsy). Thirty seven percent of those were for HCC.
* EM navigation and fusion of real-time images with pre-acquired scans has been used in hepatic biopsies at the NIH for more than 15 years. NIH / NCI clinical trials have performed fusion biopsies with EM tracking in > 2000 patients, > 40,000 biopsies over the past 12 years.
* Indocyanine green (ICG) is an FDA approved optical molecular imaging fluorescent dye used for visualization of cells and tissues. ICG has been used for decades in ophthalmology for imaging retinal blood vessels. ICG was FDA cleared in 1959 and has been widely used to assess liver function perioperatively. ICG is administered as an injection. Adverse effects are rare and most often minor.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order be eligible to participate in this study, an individual must meet all of the following criteria:

* Patients must have imaging findings consistent with hepatocellular carcinoma or other liver neoplasms or metastasis, for whom image-guided percutaneous biopsy is planned as clinically indicated or Institutional Review Board (IRB)-approved under a separate research protocol.
* Patients must have at least one lesion that can readily be biopsied per Principal Investigator.
* Age >18 years.
* Patients must have the ability to understand and the willingness to sign a written informed consent document.
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they verbally report amenorrhea for 12 months without an alternative medical cause, or have had surgery or received chemicals to induce menopause.

EXCLUSION CRITERIA:

* History of hypersensitivity reactions to Indocyanine Green (ICG), iodinated contrast, or sulfur-containing compounds.
* Pregnant women and nursing mothers are excluded from this study because of exposure to radiation from CT scanning associated with the biopsy
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, or psychiatric illness/social situations that, in the opinion of the Principal Investigator, would limit compliance with study requirements

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-01-27 (Actual); Primary Completion 2025-01-29 (Actual); Study Completion 2025-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Pinto, M.D., Principal Investigator — National Institutes of Health National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified human data generated in this research for future research may be shared.
Time Frame: Two years after completion of study
Access Criteria: De-identified data may be shared with the following:
  * In an NIH-funded or approved public repository, www.clinicaltrials.gov.
  * In Biomedical Translational Research Information System (BTRIS)
  * In publication and/ or public presentations at the time of publication or shortly thereafter

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-CC-0039.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Optical Plus Fusion for Liver Biopsy
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Optical Plus Fusion for Liver Biopsy
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 1
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Secondary Outcome: Concordance With the Histopathology and Indocyanine Green (ICG) Fluorescent Signal at the In-vivo Site of Biopsy Using a Combination of OMI and EM Tracking
Description: The concordance with the histopathology and indocyanine green (ICG) fluorescent signal at the in-vivo site of biopsy using a combination of a handheld optical molecular imaging (OMI) and electromagnetic (EM) tracking and the target to background ratio (TBR) was obtained. Concordance is defined as a TBR ≥ 2. TBR is calculated by dividing the mean fluorescence intensity within the lesion by the mean fluorescence intensity within the adjacent liver parenchyma. Analysis was done as the median of all positive TBR readings.
Time Frame: Within 15 minutes from start of procedure
Population: All participants who completed the study and was TBR positive.
Measure: Median (Full Range); unit: Ratio
Arm/Group | Optical Plus Fusion for Liver Biopsy
Number analyzed (Participants) | 6
Ratio | 3.29 [2.47 to 35.96]

2. Secondary Outcome: Participants With Concordance Between Histopathology Outcomes and Target to Background Ratio (TBR) Using ex Vivo Fluorescence Assessment
Description: Number of participants whose ex vivo fluorescence assessment of biopsy cores obtained from the target lesion is in concordance with the histopathology result from the same cores. The point-of-care device camera was used to confirmed the presence or absence of ICG emission in biopsy cores from all patients.
Time Frame: Within 15 minutes from start of procedure
Population: All participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Optical Plus Fusion for Liver Biopsy
Number analyzed (Participants) | 7
Participants
  Positive | 6
  Negative | 1

3. Primary Outcome: Participants With Detectable Indocyanine Green (ICG) Fluorescent Signal at the In-vivo Site of Biopsy
Description: Number of Participants with detectable indocyanine green (ICG) fluorescent signal at the in-vivo site of biopsy using a combination of optical molecular imaging (OMI) and electromagnetic (EM) tracking. Real-time EM navigation effectively guided the needle to the vicinity of the target lesion, allowing subsequent OMI to be performed to provide in situ confirmation of ICG presence.
Time Frame: Within 15 minutes from start of procedure
Population: All participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Optical Plus Fusion for Liver Biopsy
Number analyzed (Participants) | 7
Participants | 7

ADVERSE EVENTS:
Time Frame: 18-24 hours before before procedure and up to three hours post procedure
Arm/Group | Optical Plus Fusion for Liver Biopsy
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 1/7
Other Adverse Events (participants affected / at risk) | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Optical Plus Fusion for Liver Biopsy (N=7)
Infusion related reaction (General disorders) | 1

LIMITATIONS AND CAVEATS:
Study was prematurely terminated due to recruitment difficulty.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-09): https://cdn.clinicaltrials.gov/large-docs/66/NCT04258566/Prot_SAP_000.pdf